CLINICAL TRIAL: NCT02529696
Title: Measuring Sedation in the Intensive Care Unit Using Wireless Accelerometers
Status: Terminated | Type: Observational
Why Stopped: Low enrollment, unable to power adequately
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1502M62761
Record Dates: First submitted 2015-08-10; First posted 2015-08-20 (Estimated); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia
Keywords: accelerometer; RASS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Medical device, accelerometer: A wrist and chest accelerometer will be worn for the duration of stay in the ICU. Data will be generated from patient movement and recorded. Neither the generated data or the worn devices will influence care team's decisions during the patients' stay.
  Interventions: Device: Accelerometer

INTERVENTIONS:
Device: Accelerometer — Measures patient movement

SUMMARY:
Maintenance of analgesia during a patient stay in the hospital has been an important area of investigation after demonstrating a direct correlation between level of sedation and mortality in the ICU setting. This study will investigate the use of accelerometers in determining patient sedation level.

DETAILED DESCRIPTION:
The goal of the study is to use accelerometers to track patient movement while under sedation in the ICU. Analysis of patient movement may reveal objective means to measuring patient level of sedation. Average length of stay is estimated to be one week.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the neuro ICU at University of Minnesota

Exclusion Criteria:

* Unable to wear accelerometer device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving care from the neuro ICU at the University of Minnesota will be eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Accelerometer movement | Duration of ICU stay: estimated to be one week
  Movement during stay in the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD/MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No